CLINICAL TRIAL: NCT00243477
Title: MOTIV Study. Effect of Antidepressive Treatment by Escitalopram Started Preoperatively in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: MOTIV Study- Effect of Antidepressive Treatment by Escitalopram in Patients Undergoing Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Jean Minjoz (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Prof. Sidney Chocron, MD,PhD, Hopital Jean Minjoz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-395
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass; Surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Escitalopram given
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo given
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10mg or placebo once a day
  Other Names: Seroplex

SUMMARY:
The purpose of this study is to determine the effect of an antidepressive medication (Escitalopram), started preoperatively and given during 6 months, on 6-month and 1 year post-operative morbidity and mortality after coronary artery bypass grafting

DETAILED DESCRIPTION:
Depression is known to have an adverse effect on post-operative mortality and morbidity after coronary artery bypass grafting. Cardiac surgery is known to cause transient depression in patients. The purpose of this double-blind, randomized study is to determine the effect of an antidepressive medication (Escitalopram), started preoperatively and given during 6 months, on 6-month and 1 year post-operative morbidity and mortality after coronary artery bypass grafting. Treatment is given from 21 to 15 days pre-operatively until the 6th post-operative month. Morbidity as defined by the STS database as well as mortality is checked during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary artery bypass surgery
* > 30 years old

Exclusion Criteria:

* Contra-indication to antidepressive treatment
* Already treated by antidepressive treatment
* Concomitant cardiac surgery as valve replacement etc.
* Patients having anticoagulation therapy
* Pregnant women
* Hepatic insufficiency

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2006-01; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Postoperative morbi-mortality | 6 months and 1 year
  (1) cardiac : (2) pulmonary (3) neurologic (4) renal (5) rythm (6) infectious(7) any surgery or invasive procedure necessary to treat a postoperative adverse event associated with the initial cardiac surgery ; (8) myocardial infarction during follow-up; (9) congestive heart failure during follow-up; (10) rehospitalization for cardiac related cause, and (11) rehospitalization for non-cardiac related cause

SECONDARY OUTCOMES:
Quality of life measured by SF-36 | preoperatively and 1,3,6, and 12 months post-operatively
  Influence of treatment on Quality of Life after surgery
Beck depression index (BDI) and Center for Epidemiologic Studies Depression (CES-D) Scale | preoperatively, and 1,3,6, and 12 months post-operatively.
  Morbi-mortaity and quality of life according to preoperative values of BDI and/or CES-D

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Chocron, Prof, Study Chair — Department of Cardiac Surgery - Besancon - France
Locations (1):
- Sidney Chocron, Besançon, Doubs, France